CLINICAL TRIAL: NCT06660459
Title: Pattern of Menorrhagic Female Attending the Hematology Unit in Assuit University Children Hospital
Acronym: Menorrhagia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hasnaa Fawzy Abdelbasir Ibrahim, Doctor, Assiut University
Other Study IDs: Menorrhagic female
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Menorrhagia
Keywords: Menorrhagia
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To Evaluate Causes of Menorrhagia in Adolescent FemalesSpecially Hematological causes to help in management of abnormal uterine bleeding.

DETAILED DESCRIPTION:
Abnormal uterine bleeding (AUB) is defined as bleeding from uterine corpus that is abnormal in duration, volume, frequency and/or regularity. Due to immaturity of the hypothalamic-pituitary-ovarian (HPO) axis, AUB is common in adolescents. [1] Furthermore, inherited or acquired bleeding disorder may further intensify the existing hormonal imbalance and increase morbidity of the underlying condition.

In addition to these problems, hyperprolactinemia, thyroid disorders and polycystic ovary syndrome (PCOS) are the common underlying endocrine disorders. [2] Abnormal Uterine Bleeding decreases quality of life, affects school attendance and limits sports and social activity participation. [3] The normal menstrual cycle depends on the feedback loops of estrogen and progesterone on the production of luteinizing hormone and follicle-stimulating hormone by the pituitary gland and on the hypothalamus's normal function as metronome for the hypothalamic-pituitary- ovarian axis. [4] Differential diagnosis of abnormal uterine bleeding in adolescents: Bleeding disorders: (Von Willebrand disease, Platelet dysfunction Thrombocytopenia, Clotting factor deficiency) Endocrine causes: (Anovulatory bleeding, Polycystic ovary syndrome, Thyroid disorders, Hyperprolactinemia ).

Gynacological causes: (Adenomyosis, leiomyoma,polyp, malignancy, ovulatory dysfunction)(5) Medications: (Anticoagulants, Depot medroxyprogesterone, implants Intrauterine devices). [7] A woman's monthly menstruation takes a large toll on the hemostatic system. To avoid excessive bleeding. Any quantitative or qualitative disruption of the hemostatic

system can lead to increased menstrual bleeding. Primary hemostasis: involves the integration of platelets and von Willebrand factor (VWF). Initiation of primary hemostasis begins with injury to the blood vessel wall.

This injury allows exposure of collagen, elastin, and VWF causes platelets to activate and bind to VWF. Platelets are activated to signal further platelet activation and aggregation , which leads to the formation of the primary hemostatic plug. [8] Secondary hemostasis involves coagulation proteins called factors, the blood vessel wall, and fibrin. Endothelial wall injury causes the release of tissue factor ,which activates factor(F)VII to the activated form, FVIIa.15 The tissue factor/FVIIa complex activates the remainder of the coagulation cascade and the formation of thrombin. The final step is the activation of FXIII ,which cross links fibrin chains to form the fibrin clot. Anticoagulants, such as protein C,S , and antithrombin, as well as plasmin, help balance this procoagulant state and prevent excessive thrombus formation. [9] Most adolescents need outpatient management and reassurance that their menstrual cycles would become cyclic and ovulatory over time. However, treatment is required when AUB causes anemia or impairs quality of life . In these girls, the first line treatment is generally medical. Acute AUB patients who are clinically unstable, have active bleeding or severe anemia should be hospitalized for management A clinical decision should be made regarding intravenous crystalloid and blood or blood product transfusions, hormone treatment, and iron replacement, according to the severity of bleeding, clinical condition of the patient, hemodynamic stability and the underlying medical problem. If an underlying cause can be identified, appropriate specific treatment should be given

ELIGIBILITY:
Inclusion Criteria:

- 1. Age of female patients range from (9 -18) years old.

2. Girls with heavy menstrual bleeding

Exclusion Criteria:

* 1. Patients on medication affecting coagulation profile. 2. Patients with pre-existing illness as chronic lung, liver, renal disease or malignancy.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Female from age 8 years to age 18 years diseased with menorrhagia and help In dignosis and prevent utrine bleeding
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Evalution Causes of Menorrhagia in Adolescent FemalesSpecially Hematological causes to help in management | Baseline
  Evalution Causes of Menorrhagia in Adolescent Females Specially Hematological causes to help in management

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] ACOG Committee Opinion No. 651: Menstruation in Girls and Adolescents: Using the Menstrual Cycle as a Vital Sign. Obstet Gynecol. 2015 Dec;126(6):e143-e146. doi: 10.1097/AOG.0000000000001215. PMID 26595586
- [Result] Barbieri RL. The endocrinology of the menstrual cycle. Methods Mol Biol. 2014;1154:145-69. doi: 10.1007/978-1-4939-0659-8_7. PMID 24782009